CLINICAL TRIAL: NCT00101842
Title: Phase I/II Study of Gemzar and Platinol Followed by Alimta and Gemzar in Patients With Advanced or Metastatic Bladder Cancer
Brief Title: Gemcitabine and Platinol Followed by Pemetrexed and Gemcitabine in Patients With Advanced or Metastatic Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9439; H3E-US-S066
Record Dates: First submitted 2005-01-14; First posted 2005-01-17 (Estimated); Last update posted 2006-08-29 (Estimated); Status verified 2006-08

CONDITIONS: Carcinoma, Transitional Cell
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Pemetrexed; Gemcitabine; Cisplatin

INTERVENTIONS:
Drug: Pemetrexed
Drug: Gemcitabine
Drug: Platinol

SUMMARY:
The purposes of this study are: To determine the maximum tolerated dose of Gemcitabine and Platinol followed by Pemetrexed and Gemcitabine in patients with advanced or metastatic transitional cell carcinoma of the urothelium; To determine the safety of Gemcitabine and Platinol followed by Pemetrexed and Gemcitabine and any side effects that might be associated with the combination of these drugs; To determine whether Gemcitabine and Platinol followed by Pemetrexed and Gemcitabine can help patients with advanced bladder cancer live longer; To determine whether Gemcitabine and Platinol followed by Pemetrexed and Gemcitabine can make your tumor smaller or disappear, and for how long.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven metastatic bladder cancer
* No prior chemotherapy for metastatic disease except before or after surgery, which was completed 6 months before enrollment
* Prior radiation allowed, if it is not the only site of measurable disease and if completed 3 weeks before enrollment
* 18 years of age and older

Exclusion Criteria:

* Pure adeno- or squamous urothelial cancer
* Brain metastases that causes symptoms
* Have not received treatment within the last 30 days with a drug that has not received regulatory approval for any indication
* Inability to take dexamethasone, folic acid or vitamin B12, according to the protocol
* Clinically relevant fluid collection in the lungs or abdomen that cannot be controlled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61
Dates: Start 2004-12; Study Completion 2006-07

PRIMARY OUTCOMES:
Toxicity will be measured by standard grading methods.

SECONDARY OUTCOMES:
Response will be measured by Response Evaluation Criteria in Solid Tumors (RECIST).
Duration of response is defined as time from first objective assessment of CR or PR to first time of progression or death from any cause.
Time to progressive disease is defined as time from enrollment to first date of disease progression.
Time to treatment failure is defined as time from enrollment to first observation of disease progression, death of any cause or early discontinuation of treatment.
Survival time is defined as time from enrollment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Dallas, Texas, United States